CLINICAL TRIAL: NCT07359807
Title: Head-to-Head Comparison of Sirolimus Versus Paclitaxel Drug-Eluting Balloon Angioplasty in the Femoropopliteal Arteries
Brief Title: A Prospective, Randomized, Multi-center Trial Comparing the MagicTouch PTA Sirolimus-coated Balloon to Paclitaxel-coated Balloons for the Treatment of Stenotic or Occluded Femoropopliteal Arteries in Peripheral Arterial Disease (PAD) Patients.
Acronym: MAGICAL SFA
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Concept Medical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CM-US-R06
Record Dates: First submitted 2026-01-21; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Popliteal Artery Disease; Superficial Femoral Artery Disease
Keywords: SFA; Sirolimus; Paclitaxel; Drug-eluting; Angioplasty; Balloon; MagicTouch; PAD; Peripheral Arterial Disease; Stenotic; Stenosis; Occlusion; Superfical Femoral Artery; Popliteal Artery
MeSH Terms: conditions — Peripheral Arterial Disease; Constriction, Pathologic; Bites and Stings | interventions — Sirolimus

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Parties will remain masked until the primary endpoint is passed. Masking will be maintained as best as can be for care providers beyond those directly responsible for the index procedure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- MagicTouch sirolimus drug coated angioplasty balloon (Experimental): Subjects randomized to this arm will receive the experimental device during the angioplasty procedure to treat the affected vessel lesion that was occluded or stenosed.
  Interventions: Combination Product: Sirolimus (RAPAMUNE) drug-coated balloon angioplasty catheter
- Paclitaxel drug coated angioplasty balloon (Active Comparator): Subjects randomized to this arm will receive the control device during the angioplasty procedure to treat the affected vessel lesion that was occluded or stenosed.
  Interventions: Combination Product: Paclitaxel drug-coated balloon angioplasty

INTERVENTIONS:
Combination Product: Sirolimus (RAPAMUNE) drug-coated balloon angioplasty catheter — Sirolimus is used outside the United States to block cell growth, cell proliferation (especially T-cells), and angiogenesis (new blood vessel formation). This experimental device uses proprietary technology to adhere sirolimus to the balloon catheter, deliver it to the affected vessel, and ultimately be absorbed by the surrounding tissue.
  Arms: MagicTouch sirolimus drug coated angioplasty balloon
Combination Product: Paclitaxel drug-coated balloon angioplasty — Paclitaxel, which is used in cancer chemotherapy for various indications, is a drug that disrupts normal microtubule function and prevents neointimal hyperplasia by inhibiting smooth muscle cell migration, proliferation, and extracellular matrix secretion and is currently used in the United States.
  Arms: Paclitaxel drug coated angioplasty balloon

SUMMARY:
Percutaneous Transluminal Angioplasty (PTA), in which a balloon is advanced and inflated in the obstructed artery for several seconds to minutes, has become the standard endovascular treatment for peripheral arteries. The long-term success of bare balloon PTA in the femoropopliteal segment is hampered by the occurrence of restenosis, which can be reduced by local antiproliferative drug delivery via the PTA balloon catheter.

The rationale of this trial is based on the hypothesis that the usage of the MagicTouch drug-coated balloon (DCB) is at least equal (non-inferior) with regard to efficacy and safety in comparison with a clinically well-established paclitaxel drug-coated balloon (PTX DCB).

The objective of this prospective, randomized, multi-center trial is to compare the Magic Touch® DCB with PTX DCBs for treatment of high-grade stenotic or occluded lesions in supeficial femoral artery (SFA) and/or P1 segment of the popliteal artery in PAD patients.

ELIGIBILITY:
Inclusion Criteria:

* Subject age ≥ 21 years
* Subject has been informed of the nature of the trial, the duration of the trial, agrees to attend follow-up visits, agrees to complete the required testing, agrees to participate, and has signed an informed consent form.
* Rutherford category 2-4 according to the investigator's subjective evaluation
* Subject has de-novo or re-stenosed lesion with ≥ 70% stenosis documented angiographically, and no prior stent in the target lesion.
* Target lesion length is ≥ 40mm and ≤ 200mm by visual estimate of the treating physician.
* Multiple lesions with max. A 30mm healthy vessel segment between lesions can be considered, at the treating physician's discretion, as one lesion. Total lesion length should not exceed 200mm.
* Reference vessel diameter (RVD) ≥ 4mm and ≤ 7 mm by visual estimation.
* Patency of P2 and P3 segments of the popliteal artery and at least one (1) infra-popliteal artery to the ankle (< 50% diameter stenosis) in continuity with the femoropopliteal artery.
* Patency of the ipsilateral iliac artery (≤ 30% diameter stenosis). Iliac artery stenosis > 30% may be treated during the index procedure to ensure sufficient inflow.
* Staged Intervention of the contralateral limb is permitted at +/- 30 days.
* A subject can only be enrolled and randomized once with only one target lesion in the MAGICAL SFA trial. Note that only the lesion in one limb can be treated as a target lesion for the index procedure.

Exclusion Criteria:

* Failure of the guidewire to successfully cross the target lesion or subintimal target lesion.
* Flow-limiting dissection after pre-dilatation and/or residual stenosis > 30% prior to randomization.
* Angiographic evidence of severe calcification of the target vessel (contiguous calcification on both sides of the vessel).
* Presence of fresh/organized thrombus in the target lesion.
* Presence of aneurysm in the target vessel/s.
* Prior vascular surgery (including atherectomy , bypass surgery) of the target limb.
* Prior stent in the target lesion.
* Stroke or heart attack within three months prior to enrollment.
* Any vascular surgical procedure or intervention performed in the target limb within 30 days prior to or planned within 30 days post index procedure.
* Any vascular treatment with PTX or sirolimus-coated devices 60 days prior to the index procedure.
* Target lesion requires treatment with alternative therapies such as primary stenting, laser, lithotripsy, thrombectomy, atherectomy, and/or cryoplasty brachytherapy re- entry devices.
* Enrolled in another investigational drug, device, or biologic trial where the primary end point is not yet achieved.
* Life expectancy of less than one year in the investigator's opinion.
* Known allergies or sensitivity to heparin, aspirin, other anticoagulant/antiplatelet therapies, sirolimus, paclitaxel, or contrast media that cannot be adequately pre- treated prior to index procedure.
* Significant gastrointestinal bleeding or any coagulopathy that would contraindicate the use of anti-platelet therapy.
* Receiving dialysis or immunosuppressant therapy . (A systemic corticosteroid therapy with expected maximum dosage of 5mg prednisolone or equivalent, per day, during the initial 9 months after procedure, is allowed.)
* Subjects with severe (Stage 4) renal disease, defined as eGFR < 30%.
* Pregnant or lactating females .
* History of major amputation in the target lesion limb.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 478 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2033-01 (Estimated)

PRIMARY OUTCOMES:
Primary Efficacy Endpoint | One year from index procedure
  The absence of clinically driven target lesion revascularization (CD-TLR) due to symptoms and drop of ABI of ≥ 20% or > 0.15 when compared to post-procedure or restenosis with PSVR > 2.4 evaluated by duplex ultrasound.

SECONDARY OUTCOMES:
Secondary Safety Endpoint | One year after index procedure
  Freedom from device and procedure-related death through 12 months post-procedure, as well as freedom from both target limb major amputation and clinically driven target vessel revascularization.

CONTACTS AND LOCATIONS:
Overall Officials: Farhana Siddique, Study Director — Concept Medical Inc.; Sahil Parikh, MD, Principal Investigator — New York-Presbyterian/Columbia University Hospital; Eric A Secemsky, MD, Principal Investigator — Beth Israel Deaconess Medical Center; Brain DeRubertis, MD, Principal Investigator — New York Presbyterian - Weill Cornell Medical Center; Edward Choke, PhD, Principal Investigator — Sengkang General Hospital; Masahiko Fujihara, MD, Principal Investigator — Kishiwada Tokushukai Hospital

IPD SHARING:
Plan to Share IPD: No
This may change, but at this time, the results are for potential future marketing and sales of the investigational device pending government approval.